CLINICAL TRIAL: NCT01396317
Title: Phase IIa of Tocilizumab In the Treatment of Polymyalgia Rheumatica
Brief Title: Study of Tocilizumab to Treat Polymyalgia Rheumatica
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11081
Record Dates: First submitted 2011-07-11; First posted 2011-07-18 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Polymyalgia Rheumatica (PMR)
Keywords: PMR; POLYMYALGIA RHEUMATICA; Tocilizumab; Hospital for Special Surgery; HSS; Robert Spiera
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tocilizumab (Experimental): This is a single-arm study. All subjects will receive the active study treatment for 12 months, and will then be evaluated for 3 months of long-term follow-up.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab is a humanized anti-interleukin-6 receptor antibody that has been FDA approved for the treatment of rheumatoid arthritis (RA). This molecule binds to the IL-6 binding site of human IL-6 receptor, and competitively inhibits IL-6 signaling.
  Other Names: Actemra

SUMMARY:
This is a fifteen-month open label, Phase IIa clinical trial is being conducted to assess the tolerability, safety and efficacy of a medication called Tocilizumab (Actemra®) in patients with polymyalgia rheumatica (PMR).

DETAILED DESCRIPTION:
This fifteen-month open label, Phase IIa clinical trial is being conducted to assess the tolerability, safety and efficacy of a medication called Tocilizumab (Actemra®) in patients with polymyalgia rheumatica (PMR). The typical symptoms of PMR are muscle pain and stiffness in the shoulder, neck or hip region. Steroids have traditionally been used to treat this condition with great success, although long courses of steroids, up to 2 years in many cases, are often required. This can result in many unwanted side effects including diabetes, high blood pressure, heart disease, cataracts, weak bones with fractures, weak muscles, skin bruising, difficulty sleeping and mood disturbances. In this trial, the steroid dosage will be decreased much more quickly than what is done in routine clinical practice; there is an expectation that steroid therapy will be withdrawn within six months.

Tocilizumab is a medication already on the market that has been FDA approved in the US and Japan for the treatment of rheumatoid arthritis, and in Japan it is also approved for certain types of juvenile idiopathic arthritis (which is like rheumatoid arthritis in children) and Castleman's disease (which is a rare disease that causes enlarged lymph nodes). It is not FDA approved to treat polymyalgia rheumatica at this time. In this study, it will be given as an intravenous infusion once a month for a treatment period of one year. Experiments done on the blood of patients with PMR show one particular cytokine or small molecule that circulates throughout the body, interleukin-6, to be elevated in this disease. Tocilizumab is a medication that is designed to specifically block this cytokine. The co-primary endpoints for this study include efficacy, as well as evaluations of safety and tolerability.

* Efficacy will be defined by the proportion of patients in Disease Remission (DR) off corticosteroids, without relapse or recurrence, at six months from trial entry
* Safety and tolerability of Tocilizumab will be evaluated during the fifteen-month study period by the monitoring of adverse events and immunogenicity surveillance

Disease Remission (DR) will be defined as the disappearance of signs and symptoms of polymyalgia rheumatica (aching and stiffness of the shoulder, hip girdle, or both) with normalization of erythrocyte sedimentation rate (ESR<30 mm/hr) and c-reactive protein (CRP ≤1.0 mg/dl), unless elevation of ESR and/or CRP are attributable to causes other than PMR (i.e., infection).

ELIGIBILITY:
Disease- Specific Inclusion Criteria:

Patients must meet the following inclusion criteria to be eligible for study entry:

Diagnosed with polymyalgia rheumatica and enrolled within one month of diagnosis.

Disease Specific Exclusion Criteria:

Patients will be excluded from the study based on the following criteria:

* Symptoms or diagnosis of temporal arteritis, including headache, jaw claudication, hyperesthesia of scalp, abnormal palpated temporal artery, visual disturbances, temporal artery biopsy positivity
* Concurrent rheumatoid arthritis
* Presence of rheumatoid factor and CCP
* Other inflammatory arthritis or other connective tissue diseases, such as but not limited to systemic lupus erythematosus, systemic sclerosis, vasculitis, polymyositis, dermatomyositis, mixed connective tissue disease
* Treatment of polymyalgia rheumatica with more than 20mg of daily prednisone or its equivalent at the time of screening
* Treatment with more than 30mg of daily prednisone or its equivalent since diagnosis. Treatment with 30mg of daily prednisone or its equivalent since diagnosis for more than 2 weeks.
* More than 4 weeks of corticosteroid therapy prior to enrollment
* History of bowel perforation within the past five years.
* Active diverticulitis.
* Pre-existing or recent onset demyelinating disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Spiera, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab + Corticosteroid Taper: In a single-center open-label study, subjects with newly diagnosed PMR (Healey criteria) and prior treatment with <1 month of corticosteroids (CS) were treated with TCZ 8mg/kg IV monthly for 12 months plus a rapid CS taper. Subjects were followed for 15 months. Those with concurrent GCA or those treated with >30mg prednisone were excluded.
- Control (Corticosteroid Taper Alone): A cohort of consecutively evaluated patients with newly diagnosed PMR who declined participation in the trial or failed to meet inclusion criteria served as a control group. These patients were treated contemporaneously by a single rheumatologist with expertise in PMR and received CS alone, tapered at the treating physician's discretion.
Period: Overall Study
Arm/Group | Tocilizumab + Corticosteroid Taper | Control (Corticosteroid Taper Alone)
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tocilizumab + Corticosteroid Taper: All subjects will receive the open-label active study treatment for 12 months, and will then be evaluated for 3 months of long-term follow-up.
  Tocilizumab: Tocilizumab is a humanized anti-interleukin-6 receptor antibody that has been FDA approved for the treatment of rheumatoid arthritis (RA). This molecule binds to the IL-6 binding site of human IL-6 receptor, and competitively inhibits IL-6 signaling.
- Control (Corticosteroid Taper Alone): A cohort of consecutively evaluated patients with newly diagnosed PMR who declined participation in the trial, or failed to meet inclusion criteria, served as a comparator group.These patients were treated contemporaneously with the comparator group by a single rheumatologist with expertise in PMR and received glucocorticoids alone, tapered at the treating physician's discretion, as is the standard of care in PMR.
- Total: Total of all reporting groups
Arm/Group | Tocilizumab + Corticosteroid Taper | Control (Corticosteroid Taper Alone) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8.5) | 72 (10.7) | 70 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in Disease Remission at Six Months From Trial Entry
Description: The co-primary endpoints for this study include efficacy:
  • Efficacy will be defined by the proportion of patients in Disease Remission (DR) off corticosteroids, without relapse or recurrence, at six months from trial entry
  Relapse was defined as the reappearance of signs and symptoms of PMR, accompanied by an increasing erythrocyte sedimentation rate and/or C-reactive protein level attributable to disease activity. Recurrence was similarly defined as the return of PMR symptoms in conjunction with elevations in levels of inflammation markers, occurring 1 month after discontinuation of glucocorticoid therapy.
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab + Corticosteroid Taper | Control (Corticosteroid Taper Alone)
Number analyzed (Participants) | 9 | 10
Participants | 9 | 0

2. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: The co-primary endpoints for this study include evaluations of safety and tolerability:
  • Safety and tolerability of Tocilizumab will be evaluated during the fifteen-month study period by the monitoring of adverse events and immunogenicity surveillance
Time Frame: 15 months
Measure: Number; unit: Number of Adverse Events
Arm/Group | Tocilizumab
Number analyzed (Participants) | 10
Number of Adverse Events
  Adverse Events | 23
  Serious Adverse Events | 1

3. Secondary Outcome: Proportion of Patients Able to Achieve Disease Remission (DR) Off Corticosteroids, Without Disease Relapse or Recurrence
Time Frame: 12 and 15 months from trial entry
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab + Corticosteroid Taper | Control (Corticosteroid Taper Alone)
Number analyzed (Participants) | 9 | 0
Participants | 9 | 0

4. Secondary Outcome: Proportion of Patients Who Develop Disease Relapses
Description: Relapse was defined as the reappearance of signs and symptoms of PMR, accompanied by an increasing erythrocyte sedimentation rate and/or C-reactive\ protein level attributable to disease activity. Recurrence was similarly defined as the return of PMR symptoms in conjunction with elevations in levels of inflammation markers, occurring 1 month after discontinuation of GC therapy.
Time Frame: 6, 12 and 15 months from trial entry
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab + Corticosteroid Taper | Control (Corticosteroid Taper Alone)
Number analyzed (Participants) | 9 | 10
Participants | 0 | 10

5. Secondary Outcome: The Cumulative Dose of Prednisone
Time Frame: 6, 12 and 15 months from trial entry
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Tocilizumab + Corticosteroid Taper | Control (Corticosteroid Taper Alone)
Number analyzed (Participants) | 9 | 10
milligrams | 1,085.3 (301.3) | 2562.0 (1355.9)

6. Secondary Outcome: Total Number of Relapses/Recurrences
Time Frame: 12 months
Measure: Number; unit: Incidents
Arm/Group | Tocilizumab + Corticosteroid Taper | Control (Corticosteroid Taper Alone)
Number analyzed (Participants) | 9 | 10
Incidents | 0 | 7

ADVERSE EVENTS:
Time Frame: 4 years
Description: Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed for the control group (corticosteroid taper alone).
Arm/Group | Tocilizumab + Corticosteroid Taper
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab + Corticosteroid Taper (N=10)
Non-displaced fracture of sternum with small anterior hematoma (Injury, poisoning and procedural complications) | 1 (1) — Car accident: Patient was seated on the passenger side of the vehicle, and was hit from the rear passenger's side and the vehicle hit the center divider. Patient was diagnosed with a non-displaced fracture of the sternum with small anterior hematoma.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab + Corticosteroid Taper (N=10)
Neutropenia (Blood and lymphatic system disorders) | 1 (7)
Viral Infection (Infections and infestations) | 1 (1)
Infusion Reaction (Injury, poisoning and procedural complications) | 1 (1) — After only receiving about 30cc of study drug during this infusion, the subject began to experience flushing and subsequently, chills. Subject was treated appropriately for the infusion reaction, and was then withdrawn from the trial.
Light-Headedness (General disorders) | 1 (1)
Nose bleeds (Blood and lymphatic system disorders) | 1 (1)
Elevated Cholesterol (Blood and lymphatic system disorders) | 1 (2)
Left Rotator cuff tendinosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sinus Infection (Infections and infestations) | 1 (1)
Trigger Finger Surgery (Surgical and medical procedures) | 1 (1)
Tricompartmental Osteoarthritis of Right Knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No